CLINICAL TRIAL: NCT05777083
Title: A Trial for the Possibility of Earlier Diagnosis of Inferior Wall ST-elevation Myocardial Infarction Using a Six-lead Handheld EKG Recorder (Kardiamobile 6L)
Brief Title: A Trial for the Earlier Diagnosis of Inferior Wall STEMI Using a Six-lead Handheld EKG Recorder
Acronym: HINT-MI
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ewha Womans University Mokdong Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: HINT-MI
Record Dates: First submitted 2023-01-19; First posted 2023-03-21 (Actual); Last update posted 2023-03-21 (Actual); Status verified 2023-03

CONDITIONS: ST Elevation Myocardial Infarction; Electrocardiogram
Keywords: Kardiamobile 6L
MeSH Terms: conditions — ST Elevation Myocardial Infarction

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Inferior STEMI group (Experimental): Patients who undergo emergent coronary angiography for ST-elevation myocardial infarction.
  Interventions: Diagnostic Test: KardiaMobile 6L
- Control group (Active Comparator): Patients who undergo elective coronary angiography to differentiate angina symptom. ST-elevation myocardial infarction will be excluded.
  Interventions: Diagnostic Test: KardiaMobile 6L

INTERVENTIONS:
Diagnostic Test: KardiaMobile 6L — Before coronary angiography, all participants will contact both fingers on the two probes at the front side of portable 6-leads electrocardiogram recorder (KardiaMobile 6L), and be recorded all six leads by contacting the other side of probe at lower extremities (left hip bone ridge, thigh, knee, lower abdomen, etc.).

SUMMARY:
The goal of this clinical trial is to compare the result from the a six-leads handheld electrocardiogram (ECG) recorder (KardiaMobile 6L) with those of the standard 12-leads ECG at the patients of acute inferior wall ST-elevation myocardial infarction (STEMI), then ultimately reduce the time it takes to perform re-through treatment according to the faster diagnosis.

Participants with STEMI who visited the emergency room will be recorded 6-leads ECG using KardiaMobile 6L in addition to the standard 12-lads ECG, which is basically performed for all patients of acute coronary syndrome.

ELIGIBILITY:
Inclusion Criteria:

* Among the patients over 19-year-old, patients of ST-elevation myocardial infarction who visit the emergency room and perform emergency coronary angiography or
* Among the patients over 19-year-old, patients who visit outpatient clinics and perform elective coronary angiography for evaluating chest pain

Exclusion Criteria:

* Patients with severe complications of myocardial infarction; cardiogenic shock, respiratory failure and mental change
* Patients who are unable to agree or disagree a written consent

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 216 (Estimated)
Dates: Start 2023-01-01 (Actual); Primary Completion 2023-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Height (amplitude) of the ST segment of lead II, III and aVF at portable 6-leads electrocardiography (ECG) from KardiaMobile 6L before coronary angiography (CAG) | pre-intervention
  Height (amplitude) of the ST segment of lead II, III and aVF at portable 6-leads ECG obtained using KardiaMobile 6L between the ER visit and performing emergent CAG (experimental group) or between the admission and elective CAG (control group).
Height (amplitude) of the ST segment of lead II, III and aVF at portable 6-leads ECG from KardiaMobile 6L after CAG | immediately after the intervention (within 30 minutes)
  Height (amplitude) of the ST segment of lead II, III and aVF at portable 6-leads ECG obtained using KardiaMobile 6L within 30 minutes of the end of the CAG.
Height (amplitude) of the ST segment of lead II, III and aVF at 6-leads ECG from monitoring equipment before CAG | pre-intervention
  Height (amplitude) of the ST segment of lead II, III and aVF at 6-leads ECG obtained from monitoring equipment at angiographic room between the time of ER visit and performing emergent CAG (experimental group) or between the admission and performing elective CAG (control group).
Height (amplitude) of the ST segment of lead II, III and aVF at 6-leads ECG from monitoring equipment after CAG | immediately after the intervention (within 30 minutes)
  Height (amplitude) of the ST segment of lead II, III and aVF at 6-leads ECG obtained from monitoring equipment at angiographic room within 30 minutes of the end of the CAG.
Height (amplitude) of the ST segment of lead II, III and aVF at Standard 12-lead ECG before CAG | pre-intervention
  Height (amplitude) of the ST segment of lead II, III and aVF at Standard 12 lead ECG which is taken between the time of ER visit and performing emergent CAG (experimental group) or between the admission and performing elective CAG (control group).
Height (amplitude) of the ST segment of lead II, III and aVF at Standard 12-lead ECG after CAG | immediately after the intervention (within 30 minutes)
  Height (amplitude) of the ST segment of lead II, III and aVF at Standard 12 lead ECG which is taken within 30 minutes of the end of the CAG.

SECONDARY OUTCOMES:
Angiographic results | during the procedure
  Angiographic results of CAG reported by interventional cardiologist who performed CAG. Result is recorded as below;
  1. Angiographical Disease Extent
     * 1) normal 2) minimal 3) 1-vessel disease 4) 2-vessel disease 5) 3-vessel disease
  2. Left Main Disease : 1) Yes 2) No
  3. LAD involvement : 1) Yes 2) No
  4. LCX involvement : 1) Yes 2) No
  5. RCA involvement : 1) Yes 2) No
  6. PCI performing : 1) Yes 2) No
  7. Revascularization segment : 1) RCA 2) LAD 3) LCX 4) LM

CONTACTS AND LOCATIONS:
Overall Officials: In Sook Kang, Study Chair — Ewha Womans University Mokdong Hospital
Locations (1):
- Ewha womans university mokdong hospital, Yangcheon, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Narasimha D, Hanna N, Beck H, Chaskes M, Glover R, Gatewood R, Bourji M, Gudleski GD, Danzer S, Curtis AB. Validation of a smartphone-based event recorder for arrhythmia detection. Pacing Clin Electrophysiol. 2018 May;41(5):487-494. doi: 10.1111/pace.13317. Epub 2018 Apr 15. PMID 29493801
- [Background] Kleiman R, Darpo B, Brown R, Rudo T, Chamoun S, Albert DE, Bos JM, Ackerman MJ. Comparison of electrocardiograms (ECG) waveforms and centralized ECG measurements between a simple 6-lead mobile ECG device and a standard 12-lead ECG. Ann Noninvasive Electrocardiol. 2021 Nov;26(6):e12872. doi: 10.1111/anec.12872. Epub 2021 Jul 19. PMID 34288227
- [Background] Mercer B, Leese L, Ahmed N, Holden AV, Tayebjee MH. A simple adaptation of a handheld ECG recorder to obtain chest lead equivalents. J Electrocardiol. 2020 Nov-Dec;63:54-56. doi: 10.1016/j.jelectrocard.2020.10.005. Epub 2020 Oct 16. PMID 33099175